CLINICAL TRIAL: NCT04097067
Title: Phase II Trial to Assess the Efficacy of Low Radiation Dose of 20 Gy for the Treatment of Marginal Zone Lymphoma or Follicular Lymphoma Stage I-II Localized in the Stomach or the Duodenum
Brief Title: ISRT 20 Gy for Indolent Localized Gastrointestinal (GI)-Lymphoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: International Lymphoma Radiation Oncology Group (ILROG) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UKM01_2019
Record Dates: First submitted 2019-09-17; First posted 2019-09-20 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Follicular Lymphoma (Gastric or Duodenal); Marginal Zone Lymphoma (Gastric or Duodenal)
Keywords: Lymphoma; Lymphoma, B-Cell, Marginal Zone; Neoplasms by Histologic Type; Neoplasms; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases; Lymphoma, B-Cell; Lymphoma, Non-Hodgkin; Lymphoma, follicular
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma; Neoplasms by Histologic Type; Neoplasms; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases; Lymphoma, B-Cell; Lymphoma, Non-Hodgkin | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (low-dose radiation therapy) (Experimental): Patients undergo low-dose radiation therapy with daily 2 Gy ad 20 Gy (ISRT with IMRT & IGRT).
  Blood draw for biomarker-analysis (at baseline visit/ after 4 Gy/ after 10 Gy / after 20 Gy RT/ at 3 and 6 months after RT)
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — Low dose radiotherapy with 20 Gy (10x2Gy)

SUMMARY:
This trial studies the effectivity of low-dose radiation therapy with 10x2Gy for the treatment of patients with stage I-II stomach or duodenal Lymphoma (Marginal Zone or Follicular)

DETAILED DESCRIPTION:
* Prove the effectiveness of 20 Gy (and non-inferiority to actually recommended 30 Gy) with respect to response rate 6 months after radiotherapy.
* Correlation of blood serum biomarker levels with lymphoma response to radiation treatment
* Recording of survival rates, quality of life (QoL), radiogenic toxicities and inflammation relevant molecules in blood serum.

Primary Objective:

Response rate 6 months after end of treatment, 4 categories according to GELA-criteria: CR (complete remission) = CR or pMRD (probable minimal residual disease), PR (partial remission) = rRD (responding residual disease), NC (no change), PD (progressive disease)

Secondary Objectives:

QoL according to EORTC (QLQ C30 and STO22). EFS=Event-free survival (time to any failure or death from any cause, patients in CR or PR), LSS=lymphoma-specific survival (time to death related to lymphoma or associated with the treatment, all patients), PFS=Progression-free survival (time to progression of lymphoma or death from any cause, all patients), OS=overall survival (time to death from any cause, all patients). Level of cytokines IL-1β, IL-4, IL-8, TNFalpha and other inflammation relevant molecules Syndecan1, MMP-2 and S100 proteins. Acute toxicities during treatment according to NCI-CTC, chronic toxicities according to NCI-CTC/ LENT-SOMA.

Monitoring of Adverse Events (AEs) and Serious Adverse Events (SAEs)

-Assessment of safety: Monitoring of Adverse Events (AEs) and Serious Adverse Events (SAEs)

ELIGIBILITY:
Inclusion Criteria:

* primary indolent gastric or duodenal lymphoma
* pathology: marginal zone lymphoma (MZL) or follicular lymphoma (FL)
* stage: clinical stage I or II (Ann Arbor classification)
* H. pylori negative or antibiotic resistant lymphoma
* IPI or FLIPI score low - high (0-4)
* any size of tumor or affected lymph nodes
* male or female with age ≥ 18 years
* performance status ECOG 0 - 3
* written informed consent by the patient

Exclusion Criteria:

* prior radiation treatment of the gastrointestinal lymphoma
* stage: clinical stage III or IV (Ann Arbor classification)-unability to understand the informed consent or unwillingness to participate in the study
* severe comorbidity or organ dysfunction contraindicating the use of RT (liver cirrhosis Child-Pugh C, chronic obstructive pulmonary disease GOLD 4, heart insufficiency NYHA IV, dialysis dependent renal insufficiency, uncontrolled epilepsy)
* known seropositivity for HIV
* acute hepatitis B or C infection
* chronic inflammatory bowel disease
* prior malignant disease (exclusion: basalioma, non-metastasized solid tumor in constant remission diagnosed >3 years ago)
* pregnancy or breastfeeding
* active substance abuse or severely compromised compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Response rate | Until 6 months after end of treatment
  4 categories according to GELA-criteria: CR (complete remission) = CR or pMRD (probable minimal residual disease), PR (partial remission) = rRD (responding residual disease), NC (no change), PD (progressive disease)

SECONDARY OUTCOMES:
QoL #1 | Until 6 months after end of treatment
  According to QLQ C30 (EORTC)
QoL #2 | Until 6 months after end of treatment
  According to STO22 (EORTC)
EFS | Until at least 6 months after end of treatment
  Event-free survival (time to any failure or death from any cause, patients in CR or PR)
LSS | Until at least 6 months after end of treatment
  Lymphoma-specific survival (time to death related to lymphoma or associated with the treatment, all patients)
PFS | Until at least 6 months after end of treatment
  Progression-free survival (time to progression of lymphoma or death from any cause, all patients)
OS | Until at least 6 months after end of treatment
  Overall survival (time to death from any cause, all patients)
Level of cytokines in blood serum | Until 6 months after end of treatment
  IL-1β, IL-4, IL-8, TNFalpha and other inflammation relevant molecules Syndecan1, MMP-2 and S100 proteins
Acute and chronic toxicities | Until at least 6 months after end of treatment
  Acute toxicities during treatment according to NCI-CTC, chronic toxicities according to NCI-CTC/ LENT-SOMA

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. H. Th. Eich, Principal Investigator — Department of Radiation Oncology University Hospital Muenster; Priv. Doz. Dr. G. Reinartz, Principal Investigator — Department of Radiation Oncology University Hospital Muenster
Locations (1):
- Department of Radiation Oncology, Münster, North Rhine-Westphalia, Germany